CLINICAL TRIAL: NCT04009941
Title: Study on the Efficacy and Safety of 4.5mg Pegylated Recombinant Human Granulocyte Colony Stimulating Factor Per Cycle in Preventing Neutropenia After Intensive Chemotherapy for Breast Cancer
Brief Title: Efficacy and Safety of 4.5mg PEG-rhG-CSF Per Cycle in Preventing Neutropenia After Intensive Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, chief of breast surgery, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BC-P26
Record Dates: First submitted 2019-06-30; First posted 2019-07-08 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Neutropenia
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEG-rhG-CSF (Experimental): Patients with breast cancer who were treated with intensive chemotherapy received PEG-rhG-CSF.
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — 4.5mg per cycle, 24 hours after chemotherapy

SUMMARY:
This is a prospective, single-center, single-arm clinical study, to evaluate the clinical efficacy, safety and tolerance of patients with early breast cancer receiving ddEC adjuvant chemotherapy, accepting PEG-rhG-CSF as primary prevention of neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients in need for adjuvant chemotherapy confirmed by histopathology, whom should accept ddEC regimen.
* ECOG<=1
* Expected survival is greater than 6 months
* Qualified for chemotherapy，WBC>=3*109/L, ANC>=1.5*109/L, Hb>=80g/L, PLT>=80*109/L. With no bleeding tendency or systemic hematology disorder symptoms.
* No obvious EKG abnormality, no obvious cardiac dysfunction, and normal left ventricular ejection fraction.
* Liver function, ALT and AST should less than 2.5 times of the upper limit.
* Renal function, Cr and BUN should less than 1.5 times of the upper limit.
* Subjects voluntarily participate in this study and sign informed consent.

Exclusion Criteria:

* Total amount of doxorubicin used in previous chemotherapy>240mg/m2, or epirubicin>360mg/m2
* Has received hematopoietic stem cell transplantation or bone marrow transplantation
* Other drugs are currently in clinical trials
* There are currently hard-to-control infections, body temperature is higher than 38 degrees.
* Received PEG-rhG-CSF treatment before enrollment
* Received chemotherapy in 4 weeks before enrollment
* Patients with any visceral metastasis
* Patients with severe heart, kidney, liver or any other important organs chronic diseases
* Patients with severe uncontrolled diabetes
* Patients with allergic diseases, or allergies to this product or other biological products derived from genetically engineered e. coli
* Suspected or real drug users, substance abusers, alcoholics
* Pregnant or lactating women
* Severe mental or neurological disorders that affect informed consent and adverse reactions described or observed

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
RDI for each EC chemotherapy | 60 days after the first chemotherapy
  Ratio of actual dose intensity to standard dose intensity
Chemotherapeutic dose adjustment due to neutropenia | 60 days after the first chemotherapy
  percentage of dose decreasing due to neutropenia
overall completion rate of chemotherapy | 60 days after the first chemotherapy
  calculate the overall chemo-completion rate among all patients

SECONDARY OUTCOMES:
Incidence of febrile neutropenia | 60 days after the first chemotherapy
Incidence of Grade 3/4 ACN reduction | 60 days after the first chemotherapy
  evaluate the incidence of Grade 3/4 absolute neutrophil count
Duration of Grade 3/4 ACN reduction | 60 days after the first chemotherapy
  observe the duration of Grade 3/4 absolute neutrophil count

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No